CLINICAL TRIAL: NCT03833986
Title: Effectiveness of Stress Management Program on Occupational Stress Among Public Health Centers Nurses in Jordan
Brief Title: The Effect of a Stress Management Program on Occupational Stress and Coping Strategies Among Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Jafar Alkhawaldeh, Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: J8754
Record Dates: First submitted 2019-02-03; First posted 2019-02-07 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Occupational Stress; Coping Skills
MeSH Terms: conditions — Occupational Stress

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stress management program (Experimental): The stress program will be delivered to experimental group in a six-sessions for two weeks, each session will take 2 hours (2 hours/six sessions /two weeks).
  Interventions: Other: Stress management program
- Control (No Intervention): There is no intervention for controlled group during workshop but they are put on a waiting-list to receive the intervention after the active treatment group does.

INTERVENTIONS:
Other: Stress management program — Nurses stress management program will be an experiential teaching program consisting of six sessions of stress management strategies for public health centers nurses. the workshop will be in a warm quite room with efficient light, temperature, and ventilation. The intervention group will receive handouts copies of the stress management program for each session at the end of the study.
  Arms: Stress management program

SUMMARY:
The present study is designed to focus on examining the effectiveness of the stress management program on occupational stress and coping strategies among public health centers nurses in Jordan.

the Specific Objectives that will guide this study are as follow:

1. To assess the level of occupational stress among Jordanian public health nurses who work in comprehensive health care centers.
2. To find out the association between nurses' occupational stress scores and their selected demographic variables.
3. To identify the sources of occupational stress encountered among public health centers nurses in the work setting.
4. To identify the types of coping strategies utilized by Jordanian nurses working in comprehensive health care centers.
5. To evaluate the effectiveness of stress management program on occupational stress mean score among experimental and control groups at baseline, post-test and at two months' follow-up assessment.
6. To evaluate the effectiveness of stress management program on coping strategies mean score among experimental and control groups at baseline, post-test and at two months' follow-up assessment.

This experimental study will examine differential changes in two dependent variables: occupational stress and coping strategies of public health nurses after participation in experiment. Experimental Group will participate in a stress management program and control group will not receive any intervention. The null hypotheses that guide this study are:

1. Null hypothesis (H0_1): There is no significant difference in occupational stress mean score between experimental and control groups at baseline, post-intervention and at two months' follow-up assessment. (µ1 = µ2).
2. Null hypothesis (H0_2): There is no significant difference in coping strategies mean score between experimental and control groups at baseline, post-intervention and at two months' follow-up assessment. (µ1 = µ2).

DETAILED DESCRIPTION:
This study aims to evaluate the effectiveness of stress management program on occupational stress and coping strategies among Jordanian public health centers nurses.

Methodology

1. Study Location:

   This study will be carried out in eight comprehensive public health centers in Amman city, Jordan.
2. Study Design:

   Single-blind, a cluster randomized controlled trial design (RCT) with two conditions (experimental versus control group) and three time points for this study; baseline test (T0), a post-test (immediately after the second day of intervention (T1), and follow-up at two months' post-intervention (T2).
3. Study Population Target population:

   All Jordanian public health centers nurses, accessible population: public health nurses who are working in comprehensive health care centers in Amman.
4. Sampling Frame:

   Sampling will be done in three stages. Stage 1: List of comprehensive centers in Amman city served as the sampling frame in the first step (N=8) and the centers' selected served as the sampling frame for the second stage.

   Stage 2: Eight centers will be assigned randomly, 4 centers will be assigned to each group (experimental and control groups).

   Stage 3: List of all nurses who are eligible in light of the criteria in each selected centers (experimental and control groups), simple randomization will be applied to select nurses from the list.
5. Sample Size Estimation:

   The following is sample size calculation formula:

   n = [ Z1-α /2 + Z1-β] ² ×2σ² [μ1-μ2] ² Design effect = 1-P (n-1) n = 79 per group n = 79×2= 158 With consideration an estimated 20% drop out of the subjects during the study, the final sample size calculation 190 with 95 subjects in each experimental and control groups.
6. Sampling Method:

   Two-stage random sampling technique will be used in the current study. Initially; the eight centers will assign a sequential number starting from 1 to 8, then each four centers will be allocated randomly using SPSS generator random sample to experimental and control group. lastly, a List of all participants per each center (experimental & control), the eligible nurses will be randomly selected by using simple random selection of participants using a generator from SPSS to provide relative equality of the groups in terms of gender, age, years of experience, and level of education.
7. Measuring Instrument:

   The self-reporting questionnaire contain of 4 parts; coding book, demographic data, Nursing Stress Scale (NSS) Questionnaire, and Brief Coping Orientations to Problems Experienced (COPE) Scale.
8. Data Collection Procedure:

Immediately after the last session of the intervention, the participants will be asked to complete the post-test questionnaires which is the same (Demographic) (NSS) and (COPE) questionnaires use at baseline assessment. Follow-up assessment will be done at two months post the intervention. Study data collection will start from 1 March 2019 to 31 June 2019. Directors of all select centers will be informed through written an introductory letter by the researcher to the director of each center. Then, the researcher request from each director of the select center to inform all nurses who meet eligibility criteria to attend a briefing session. A participant who agrees to participate in this study will be given a packet that includes Code book, structured demographics information form, (NSS), (COPE) questionnaires and the contact card in the Arabic language. Each questionnaire packet will be assigned a code number (3-digit code) for data analysis purpose and confidentiality (i.e. Code: I-A-1 means intervention group, center code: A and participant No: 1). Also, each participant will be given 15-30 minutes to complete the questionnaires and return to the researcher on the same day, the researcher will be revised if there any incomplete answers with the nurses and will be asked to complete them. At baseline using demographic data form, (NSS) and (COPE) questionnaires for all participants at the initial meeting, as well as (NSS), and (COPE) questionnaires immediately after the last session of intervention. Also, follow-up the study will be assessed at two months' post-intervention using (NSS) and (COPE) questionnaires.

9. Attrition prevention techniques:

1. Accurate contact information of each participant will be kept separately from the questionnaire in coding book (participant's name, phone number, and E-mail address).
2. Participants will be reminded regularly via phones or email, to fill out the questionnaire and to attend stress management program sessions whenever they have time to do so.
3. the researcher's contact information will be disclosed to each participant via card to enable participants to ask any question regarding the study during the collection period of data.

10. stress management program: Stress Program Materials a stress management program is adapted and developed with reference to effectiveness of the existing stress management program for nurses . Also, the program is designed according to the theory of stress and coping and rational emotive behavior theory. The contents of the program will deliver through the use interactive learning methods which are enjoyable, fun, and engaging.

11. Implementation of Educational Program: The stress program will be delivered to experimental group in a six-sessions for two weeks, each session will take 2 hours (2 hours/six sessions /two weeks), the day and time of stress management workshop will be arranged with nursing manager of comprehensive health care center depending on staff availability and venue for sessions, but the workshop will be in a warm quite room with efficient light, temperature, and ventilation. There is no intervention for controlled group during workshop but they are put on a waiting-list to receive the intervention after the active treatment group does. The intervention group will receive handouts copies of the stress management program for each session at the end of the study. A certificate of appreciation will be given to participants in both groups after completing the study. Nurses stress management program will be an experiential teaching program consisting of six sessions of stress management strategies for public health centers nurses. Sessions will be as follows: Session one: overview of stress (definition, causes, effects of social and occupational life, stress management styles and techniques), Session two: relaxation technique training (deep breathing exercise and progressive relaxation techniques), Session three: cognitive restructuring, which include positive self-talk and problem solving techniques, Session four: humor therapy, this session will be focusing on practicing humor through several ways (laughter videos, laughter meditation, sharing of personal anecdotes and jokes, sharing of happiness thoughts) ,Session five: time management, and Session six: assertiveness training. The validity content of those sessions will be approved from three lecturers in of the faculty medicine and health sciences -UPM and three lecturers who are specialized in mental and psychiatric health nursing teaching in two Jordanian universities. Pilot study will be conducted on a sample of 5% Jordanian public health nurses with high levels of occupational stress who will not be involved in the current study to check about the face validity of stress program.

12. Evaluation of Educational Program: Immediately after the last session of the intervention, the participants will ask to complete the post-test questionnaires which is the same (NSS) and (COPE) questionnaires use at baseline assessment. Follow-up assessment will be done at two months post the intervention.12.

13. Planning for Data Analysis : Both descriptive and inferential statistics will be used to answer the research questions of this study. The computer program, The Statistical Package for the Social Sciences (SPSS 22) will be used to describe variables of the study (Demographic data, Occupational stress, and coping strategies,). Exploratory data analysis (EDA) will be carried out to determine the normality of data. Normality will be checked using Skewness and Kurtosis as well as Smirnov-Kolmogrov tests. Equality of variances will be checked for all variables using Levine's test. Categorical variables will be analyzed for frequencies and percentages, while Continuous variables will be described using the central tendency measures (means, and medians), the dispersion measures (standard deviation), and interpercentile measures (P25, P50, and P75). Descriptive analysis of mean, median, SD, frequencies, percentages, and range will be used to describe the socio-demographic variables among Jordanian public health nurses. Independent-t test will be used to compare the study's variables at baseline between two groups.in addition paired-sample t test and repeated-measures analysis of variance (ANOVA) will be used to assess the effectiveness of the intervention on the main outcome measures over time, both within and between study groups after assessing the basic assumptions of the parametric tests; linearity, independence, homoscedasticity, and normality. The level of significance will be set at p≤0.05 and the power will be set at 80% e for statistical tests analysis. Perceived stress and coping strategies need to be statistically significant for the null hypotheses to be rejected.

14. Ethical Consideration: The study will be approved by the Ethical Committee of the Faculty of Medicine and Health Sciences / University Putra Malaysia. The study will be obtained approval from Human Research Ethics Committee / Jordanian Ministry of health. Information sheet and informed consent will be given to participants. Participants will be informed that their participation is voluntary. confidentiality for participants will be assured through coded numerically of the questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* nurses who have full-time working employment and agreed to participate in the study (by consent form).
* have more than one year of experience community care .
* Do not have any psychiatric or physical health problems.
* Do not work on fixed shift as nurses on the fixed shifts experienced higher levels of stress than the nurses on the rotating shifts (Tajvar et al., 2015)..
* Nurses had undergone stress management courses.
* Less than one year of experience in community care.
* Nurses who work in more than one center.

Exclusion Criteria:

* Nurses had undergone stress management courses.
* Less than one year of experience in community care.
* Nurses who work in more than one center.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 170 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Occupational stress will be measured by Nursing stress scale (NSS) "change is being assessed" | Occupational stress will be measured to assess the change between pre-test and up to 2 months post-test
  Nursing Stress Scale (NSS) will be used in the study to measure nurses occupational stress. it consists of 34 items distributed in 7 subscales which are: Death and Dying patients (7 items), conflict with Physicians (5 items), inadequate emotional preparation (3 items), lack of support (3 items), conflict with other nurses (5 items), work Load (6 items), and uncertainty concerning treatment (5 items). A 4-point Likert scale used to indicate the frequency of work stressors experienced by nurses from never stressful (1), to occasionally (2), to frequently (3), to very frequently stressful (4). The original scale has been reported to have high reliability as evidenced by Cronbach's coefﬁcient alpha of 0.89 for the total score, Individual subscales reliability ranged from α=0.79 to α=0.89. The NSS total scores ranging from 34 to 136, A higher score indicates a higher frequency of work stressors experienced by the participants.
coping skills will be measured by The Brief Coping Orientations to Problems Experienced (COPE) Scale "change is being assesses" | Coping strategies will be measured to assess the change between pre-test- and up to 2 months post-test
  Coping skills will be assessed by the Brief Coping Orientations to Problems Experienced (COPE) Scale, this instrument contains 28 items and has 14 sub-scales (2 items per subscale) that capture 14 ways of various coping behaviors. Each item of this instrument is endorsed by participants using a 4-point Likert scale, which ranges from 1 (I have not been doing this at all), 2 (I have been doing this a little bit), 3 (I have been doing this a medium amount), 4 (I have been doing this a lot). Total scores for each subscale will be calculated, and higher total subscale scores indicate greater perceived use of a corresponding coping behavior. Carver reported good reliability and validity with Cronbach alpha ranging from 0.50-0.90 for its subscales, demonstrating acceptable internal consistency for this instrument.

CONTACTS AND LOCATIONS:
Overall Officials: Ja'far Alkhawaldeh, PhD student, Principal Investigator — University Putra Malaysia
Locations (1):
- Ministry of Health, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alkhawaldeh JM, Soh KL, Mukhtar F, Peng OC, Alkhawaldeh HM, Al-Amer R, Anshasi HA. Stress management training program for stress reduction and coping improvement in public health nurses: A randomized controlled trial. J Adv Nurs. 2020 Nov;76(11):3123-3135. doi: 10.1111/jan.14506. Epub 2020 Aug 28. PMID 32856353